CLINICAL TRIAL: NCT07208955
Title: The Effect of Heat Application and Abdominal Massage in the Early Postoperative Period on the Gastrointestinal System and Mental Well-being of Patients With Hip Fractures
Brief Title: The Effect of Heat Application and Abdominal Massage on the Gastrointestinal System and Mental Well-being of Patients With Hip Fractures
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Acelya Turkmen, Assistant Professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 151
Record Dates: First submitted 2025-09-09; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Function; Mental Well-being
Keywords: abdominal massage; gastrointestinal function; mental well-being
MeSH Terms: conditions — Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Heat application group (Experimental): The experimental group will receive heat application
  Interventions: Procedure: heat application
- Massage group (Experimental): The massage group will receive abdominal massage.
  Interventions: Procedure: abdominal massage
- placebo group (Placebo Comparator): No intervention will be performed on the placebo group.
  Interventions: Other: control group

INTERVENTIONS:
Procedure: heat application — Heat application in the early postoperative period affects gastrointestinal function and mental well-being
  Arms: Heat application group
Procedure: abdominal massage — Abdominal massage administered in the early postoperative period has an effect on gastrointestinal function and mental well-being.
  Arms: Massage group
Other: control group — control group
  Arms: placebo group

SUMMARY:
This randomised controlled trial was designed to determine the effect of early-stage heat application and abdominal massage on patients' gastrointestinal function and mental well-being following hip fracture surgery.

The study's hypotheses are as follows:

H0: Heat application and abdominal massage administered in the early postoperative period have no effect on gastrointestinal function or mental well-being.

H1: Heat application in the early postoperative period affects gastrointestinal function and mental well-being.

H2: Abdominal massage administered in the early postoperative period has an effect on gastrointestinal function and mental well-being.

The Patient Information Form, Gastrointestinal Symptom Rating Scale (GSRS) and Warwick-Edinburgh Mental Well-being Scale will be administered. Starting from the morning of the first day after surgery, patients will receive abdominal massage and heat application twice daily, in the morning and evening, for three days. The warm compress and abdominal massage will be performed consecutively. The total application time will be 30 minutes, consisting of 15 minutes of warm compress and 15 minutes of abdominal massage. Abdominal massage will be performed on patients in the experimental group using the 'abdominal massage application guidelines'. Abdominal massage involves techniques such as effleurage (stroking and spreading), petrissage (kneading) and vibration. After each application of massage, the patient's bowel sounds and movements will be listened to using a stethoscope. Before applying heat and performing the abdominal massage, care will be taken to ensure that the patient does not need to urinate, and that the room is quiet and at a suitable temperature. Patients in the experimental group will not be given laxatives, suppositories or enemas for three days; only heat application and massage will be performed during this period. During this period, researchers will assess the defecation of patients using the Bristol Stool Scale. At the end of the three-day follow-up period, patients will be asked to complete the Bristol Stool Scale, the Gastrointestinal Symptom Rating Scale and the Warwick-Edinburgh Mental Well-being Scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older,
* conscious and cooperative, with vital signs within normal limits after surgery,
* who have not defecated after surgery,
* who are able to eat orally, and
* who have a hip fracture will be included in the study.

Exclusion Criteria:

* Patients with a history of cancer, abdominal injury, delirium, or requiring intensive care will be excluded from the study.

Max Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
abdominal massage | 30 minutes
  Assessment of bowel sounds, first flatus and time of defecation.
heat application | 30 minutes
  Assessment of bowel sounds using a stethoscope

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova University, Adana, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No